CLINICAL TRIAL: NCT04636307
Title: Characterization of Retinal Disease Progression in Eyes With Non Proliferative Diabetic Retinopathy (NPDR) in Diabetes Type 2 Using Non-invasive Procedures (CHART)
Brief Title: Characterization of Retinal Disease Progression in Eyes With Non Proliferative Diabetic Retinopathy in Diabetes Type 2 Using Non-invasive Procedures (CHART)
Acronym: CHART
Status: Completed | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Collaborators: European Vision Institute Clinical Research Network (Network)
Responsible Party: Sponsor
Other Study IDs: ECR-RET-2020-15
Record Dates: First submitted 2020-10-29; First posted 2020-11-19 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: NPDR - Non Proliferative Diabetic Retinopathy; Diabetes Mellitus, Type 2; Retinal Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Retinal Diseases | interventions — Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biomarkers — To identify biomarkers obtained using non-invasive procedures that can predict disease progression and progression to sight-threatening stages of the disease and to characterize the retinal changes that occur in NPDR.

SUMMARY:
To identify biomarkers, obtained using non-invasive procedures, that can predict disease progression and progression to sight-threatening stages of the disease and to characterize the retinal changes that occur in Non Proliferative Diabetic Retinopathy (NPDR).

DETAILED DESCRIPTION:
The progression of diabetic retinopathy (DR) varies between different patients, even with similar metabolic control. It is becoming clear that a sizeable proportion of patients with mild non-proliferative diabetic retinopathy (NPDR) will take a long time to develop any sight-threatening complication. The inclusion of eyes/patients in a clinical trial that do not show any significant worsening during the period of the trial masks any beneficial effect of the drug being tested and consequently would increase trial sizes as the true therapeutic effect in high-risk patients would be partially obscured. It appears that the only option is to identify the eyes/patients that show progression of retinopathy during a pre-trial run-in period and only include such patients. Characterization of progressors in the early stages of DR and identification of biomarkers of disease progression are of major interest to facilitate drug development in this area of high unmet need.

Three different phenotypes of mild NPDR progression with different risks for development of Clinically Significant Macular Edema (CSME) were identified using cluster analysis based on the turnover rate of microaneurysms (MAT) and the central retinal thickness (CRT). Phenotype A, patients with low MAT and CRT < 260 micron in women and < 275 micron in men (on Cirrus Optical Coherence Tomography - OCT, corresponding to the mean CRT in healthy subjects plus 1 standard deviation, SD); Phenotype B, patients with low MAT and CRT ≥ 260 micron in women and ≥ 275 micron in men; and Phenotype C patients with high MAT. These phenotypes were recently confirmed in a larger population of NPDR patients. In this study, Phenotype B shows a risk for DR progression to Macular Edema (ME) of OR=13.30 and Phenotype C of OR=6.32. When CRT increase is present, then Phenotype C shows a higher risk for ME (OR=29.02). In these studies, the occurrence of proliferative diabetic retinopathy (PDR) as an outcome was rare and did not allow statistical analysis. More recently it was shown that phenotype C identifies eyes at higher risk for development of CSME and PDR, whereas phenotype A identifies eyes at very low risk for vision-threatening complications.

Patients with phenotypes B and C are, therefore, the NPDR patients with higher risk for ME development and are those patients who may benefit from early therapeutic or preventive treatment. Therefore, a proper characterization of this population is of major interest for the understanding of the disease, and to the design of new therapeutical approaches that can facilitate adequate and timely interventions.

To better characterize these patients, new non-invasive methods are now available that allow for a better insight of the retinal changes that occurs in these patients. The Optical Coherence Tomography Angiography (OCT-A) and OCT-Leakage (OCT-L) are two of these methods that can be used in longitudinal studies. These methods allow to quantify capillary closure and leakage, the main alterations occurring in DR (ischemia and leakage) and which are considered to predict sight-threatening complications, ME and PDR. In recent studies it was shown that the vessel density in the superficial and deep layers, obtained with OCT-A, and the Low Optical Reflectivity (LOR) ratio obtained with OCT-L are altered even in the earlier stages of DR. These two methods are therefore expected to better characterize leaky and ischemic patients' phenotypes (i.e., phenotypes B and C, respectively), being therefore a major step in early diagnosis and timely treatment of DR patients. Measurement of neurodegeneration (ND) represented by thinning of Ganglion Cell Layer (GCL) and Inner Plexiform Layer (IPL) will also be performed.

This study aims to better characterize the retinal changes that occur during a 2-years follow-up period in patients with diabetes Type 2 and with the initial stages of NPDR and at higher risk for sight-threatening complications, allowing better characterization of eyes at risk of progression (phenotypes B and C). The inclusion will be based on patients with established retinopathy ETDRS 35, 43, 47 and 53, distributed to the different clinical sites in the study, creating the opportunity to demonstrate the progression phenotypes.

ELIGIBILITY:
INCLUSION CRITERIA

* Diabetes type 2 according to 1985 WHO criteria;
* Age between 35 and 90 years;
* NPDR levels 35, 43, 47 or 53 (based on the ETDRS criteria - 7 fields CFP) after confirmation by the Reading Centre;
* Refraction with a spherical equivalent less than 5 Dp;
* Informed consent.

EXCLUSION CRITERIA

* Repeated HbA1C > 10% in the first visit;
* Cataract or other eye disease that may interfere with fundus examinations;
* Age-related macular degeneration, glaucoma, vitreomacular disease, or other retinal vascular disease, or any ocular condition that, in the opinion of the investigator may affect retinopathy status or alter visual acuity during the study;
* Any eye surgery within a period of 6-months;
* Previous laser treatment or previous intravitreal injections;
* Any patient comorbidity likely to affect the eye and not related with diabetes or cardiovascular disease;
* Presence of CIME (CRT ≥ 290 μm in women and ≥ 305 μm in men) with vision loss or needing immediate treatment, according to clinical practice;
* Dilatation of the pupil < 5 mm;
* Uncontrolled systemic hypertension (values outside normal range: systolic 70-210 mmHg and diastolic 50-120 mmHg).

Ages: 35 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Diabetes Type-2 and NPDR (levels 35, 43, 47 or 53)
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
DRSS severity progression | 36 months
  DRSS severity progression of one, two or more ETDRS step changes
Progression to vision-threatening complications | 36 months
  CIME defined as eyes with a CRT ≥ 290 μm in women and ≥ 305 μm in men (Zeiss Cirrus SD-OCT); CSME identified on clinical evaluation as defined by ETDRS by retinal thickening within 500 μm of the center of the fovea or presence of hard exudates (with thickening of the adjacent retina) within 500 μm of the center of the fovea, or thickening of at least 1 disc area located less than 1 disc diameter from the center of the fovea. (Zeiss Cirrus SD-OCT); PDR identified by the presence of abnormal new vessels in the retina.
Presence of ischemia | 36 months
  dentified by decrease of 2 or more Standard deviations (in relation to healthy control population) on the values of vessel density, perfusion density or FAZ circularity.

CONTACTS AND LOCATIONS:
Locations (5):
- CS042 - Department of Ophthalmology, University Hospital, CHU Dijon, Dijon, France
- Italy (3):
  - CS067- Department of Ophthalmology, University Vita Salute - Scientific Institute of San Raffael, Milan, Milan
  - CS063 - Excellence Eye Research Centre, University G. d'Annunzio of Chieti-Pescara, Pescara
  - CS020 - G. B. Bietti Eye Foundation - IRCCS, Roma
- CS001 Centre for Clinical Trials - AIBILI, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Marques IP, Reste-Ferreira D, Santos T, Mendes L, Rocha AC, Bandello F, Parravano M, Mastropasqua L, Creuzot-Garcher C, Leal S, Baschiera F, Cunha-Vaz J. One-Year Progression of Capillary Nonperfusion in Nonproliferative Diabetic Retinopathy Using Noninvasive Imaging: The CHART Study. Transl Vis Sci Technol. 2026 Jan 5;15(1):26. doi: 10.1167/tvst.15.1.26. PMID 41569021